CLINICAL TRIAL: NCT02246231
Title: The Effect of Changes in Head Position on Magnetic Resonance Image Distortion in Patients With Auditory Implants
Brief Title: Effect of Implant Position on Magnetic Resonance Image Distortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R01623
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Neurofibromatosis Type 2
MeSH Terms: conditions — Neurofibromatosis 2 | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NF2 who has an auditory implant (Experimental)
  Interventions: Device: MR imaging

INTERVENTIONS:
Device: MR imaging

SUMMARY:
Patients with Neurofibromatosis type 2 (NF2) almost always develop acoustic neuromas in both ears. As a result of the tumours themselves or the treatment of the tumours, many patients become profoundly deaf in both ears. It is possible to restore a degree of hearing by placing a hearing implant in the brainstem adjacent to the hearing pathways within the brain. This is termed an auditory brainstem implant (ABI).

The aim of this study is to find the optimum head position in relation to the MRI magnet field, which would produce least area of image distortion in patients with ABIs. This will be of benefit in optimising the MR imaging in future patients with implants.

DETAILED DESCRIPTION:
Auditory brainstem implants (ABI) are placed against the auditory centres in the brainstem if it is not possible to implant the cochlea or if the cochlear nerve, which conveys neural signals from the cochlea to the brainstem, is damaged or absent. The latter device is usually used in patients with Neurofibromatosis type 2 (NF2) who develop bilateral benign inner ear tumours called vestibular schwannomas as well as other neurological tumours1. These patients often become bilaterally profoundly deaf either as a result of the disease or because of surgery to remove the tumours and require an ABI.

Patients with NF2 require monitoring of their tumours. In the absence of an auditory implant it is possible to use magnetic resonance imaging. This is the gold standard imaging technique as it gives excellent views of the soft tissues of head. However, there has been concern regarding the use of MRI in patients with auditory implants until recently because of potential problems such as demagnetisation of the magnet within the implant, implant magnet displacement and risk to the integrity of the implant electronics. In addition, the magnet field of the implant magnet results in imaging artefact (manifesting as a signal void) around the implant site that limits the information that can be obtained.

ELIGIBILITY:
Inclusion Criteria:

- Any patient over the age of 18 with NF2 who has an auditory implant (cochlear or auditory brainstem implant) in situ and requires MRI scanning.

Exclusion Criteria:

Children under the age of 18 years Claustrophobia Bilateral implants

Contraindications and relative contraindications for MRI (as per the Radiology Department MRI protocol) including:

Pacemaker Certain metallic heart valves Ferromagnetic implanted materials and foreign bodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
To study the effect of magnet orientation in auditory brainstem implants/ cochlear implants in determining the size of signal void seen on MRI scanning. | 1 year

SECONDARY OUTCOMES:
To identify if there is an angle at which the signal void is minimised | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lloyd, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, Manchester (Manchester Borough), United Kingdom